CLINICAL TRIAL: NCT05200533
Title: Task-sharing and Shifting Model Between Family Physicians and Physiotherapists for Acute Low Back Pain Patients: a Pragmatic Cluster Randomized Controlled Trial
Brief Title: Task-sharing and Shifting Model for Acute Low Back Pain
Acronym: LombalgIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC21.0259
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Low Back Pain
Keywords: Task-sharing; Task-shifting; Family physician; Physiotherapist
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapists

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Masking Description: Data analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-sharing and shifting (Experimental): In the task-sharing and shifting group, family physicians shifted acute low back pain consultations to physiotherapists. Patients with acute low back pain are seen by the physiotherapist instead of family physician. Physiotherapist diagnose acute low back pain, identify red and yellow flags, prescribe sick leave and medications and can refer the patient to additional physical therapy treatment.
  Interventions: Other: Task-sharing and shifting model between family physicians and physiotherapists
- Usual care (Active Comparator): In the usual care group, patients with acute low back pain are seen by their family physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Task-sharing and shifting model between family physicians and physiotherapists — Medical consultations for acute low back pain patients are shifted from family physicians to physiotherapists.
  Arms: Task-sharing and shifting
Other: Usual care — Medical consultations for acute low back pain patients are performed by family physicians
  Arms: Usual care

SUMMARY:
Background: The aging population and the rising prevalence of musculoskeletal disorders increase resort to primary care services. Models of care integrating task sharing and shifting (TS/S) can help face challenge of access to care by strengthening the role of healthcare professionals. In France, a new TS/S model is being implemented between family physicians (FPs) and physiotherapists (PTs) for acute low back pain (LBP) patients' care. The aim of this study is to evaluate the effect of this new model of care on patient clinical outcomes, healthcare resources use and patient satisfaction.

Design: Pragmatic cluster randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Patients from 20 to 55 years old
* Suffering from acute low back pain since less than 4 weeks
* Able to understand and speak French
* Whose family physician is included in the task-sharing and shifting model (only in the intervention group)

Exclusion Criteria:

* Protected patient according to the public health regulation,
* Patient unable to fill the survey,
* Non-availability of the physiotherapist to receive the patient (only in the intervention group)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Effect of the TS/S model on acute low back pain (LBP) patients' disability at 6 weeks | 6 weeks after the initial consultation
  Rolland Morris Disability Questionnaire It is a 24 points scale. The lower score is 0, the higher score is 24. Higher scores mean worse outcomes as the disability level is higher.

SECONDARY OUTCOMES:
Effect of the TS/S model on acute LBP patients' disability at 3 months | 3 months after the initial consultation
  Rolland Morris Disability Questionnaire It is a 24 points scale. Scores rank form 0 to 24. Higher scores mean worse outcomes as the disability level is higher.
Effect of the TS/S model on acute LBP patient's pain at 6 weeks and 3 months | 6 weeks and 3 months after the initial consultation
  Brief Pain Inventory It is a 10 points scale. Scores rank from 0 to 10. Higher scores mean worse outcomes, as the pain level is higher.
Effect of the TS/S model on acute LBP patient's psychosocial risk factors at 6 weeks and 3 months | 6 weeks and 3 months after the initial consultation
  Start-Back screening tool It is a 9 points scale. Scores rank from 0 to 9. Higher scores mean worse outcomes.
Effect of the TS/S model on acute LBP patient's satisfaction | Few minutes after the initial consultation (less than one hour)
  Medrisk questionnaire It is a 5 points scale. Scores rank from 0 to 5. Higher scores mean better outcomes;
Effect of the TS/S model on acute LBP patient's wait time before the initial consultation | Initial consultation
  Time (number of days and hours)
Effect of the TS/S model on healthcare resources use | Initial consultation, 6 weeks and 3 months after the initial consultation
  Initial prescription of sick leave and medications, number of family physician visits, number of physical therapy appointments, number of emergency department visits at 6 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Pinsault, PhD, Study Director — University Grenoble Alps
Locations (6):
- France (6):
  - Maison de santé pluriprofessionnelle de Cran Gévrier, Annecy, Auvergne-Rhône-Alpes
  - Maison de santé pluriprofessionnelle des Hauts de Chambéry, Chambéry, Auvergne-Rhône-Alpes
  - Maison de santé pluriprofessionnelle de Voiron-Sud, Coublevie, Auvergne-Rhône-Alpes
  - Maison de santé pluriprofessionnelle de Lans-en-Vercors - Pôle Santé en Vercors, Lans-en-Vercors, Auvergne-Rhône-Alpes
  - Maison de santé pluriprofessionnelle de Moirans, Moirans, Auvergne-Rhône-Alpes
  - Pôle de santé interprofessionnel de Saint-Martin d'Hères, Saint-Martin-d'Hères, Auvergne-Rhône-Alpes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babatunde OO, Bishop A, Cottrell E, Jordan JL, Corp N, Humphries K, Hadley-Barrows T, Huntley AL, van der Windt DA. A systematic review and evidence synthesis of non-medical triage, self-referral and direct access services for patients with musculoskeletal pain. PLoS One. 2020 Jul 6;15(7):e0235364. doi: 10.1371/journal.pone.0235364. eCollection 2020. PMID 32628696
- [Background] Demont A, Bourmaud A, Kechichian A, Desmeules F. The impact of direct access physiotherapy compared to primary care physician led usual care for patients with musculoskeletal disorders: a systematic review of the literature. Disabil Rehabil. 2021 Jun;43(12):1637-1648. doi: 10.1080/09638288.2019.1674388. Epub 2019 Oct 11. PMID 31603709
- [Background] Chiarotto A, Maxwell LJ, Terwee CB, Wells GA, Tugwell P, Ostelo RW. Roland-Morris Disability Questionnaire and Oswestry Disability Index: Which Has Better Measurement Properties for Measuring Physical Functioning in Nonspecific Low Back Pain? Systematic Review and Meta-Analysis. Phys Ther. 2016 Oct;96(10):1620-1637. doi: 10.2522/ptj.20150420. Epub 2016 Apr 14. PMID 27081203
- [Background] Desmeules F, Roy JS, MacDermid JC, Champagne F, Hinse O, Woodhouse LJ. Advanced practice physiotherapy in patients with musculoskeletal disorders: a systematic review. BMC Musculoskelet Disord. 2012 Jun 21;13:107. doi: 10.1186/1471-2474-13-107. PMID 22716771
- [Background] Hill JC, Whitehurst DG, Lewis M, Bryan S, Dunn KM, Foster NE, Konstantinou K, Main CJ, Mason E, Somerville S, Sowden G, Vohora K, Hay EM. Comparison of stratified primary care management for low back pain with current best practice (STarT Back): a randomised controlled trial. Lancet. 2011 Oct 29;378(9802):1560-71. doi: 10.1016/S0140-6736(11)60937-9. Epub 2011 Sep 28. PMID 21963002
- [Background] Kechichian A, Lafrance S, Matifat E, Dube F, Lussier D, Benhaim P, Perreault K, Filiatrault J, Rainville P, Higgins J, Rousseau J, Masse J, Desmeules F. Multimodal Interventions Including Rehabilitation Exercise for Older Adults With Chronic Musculoskeletal Pain: A Systematic Review and Meta-analyses of Randomized Controlled Trials. J Geriatr Phys Ther. 2022 Jan-Mar 01;45(1):34-49. doi: 10.1519/JPT.0000000000000279. PMID 34928239
- [Derived] Kechichian A, Desmeules F, Girard P, Terrisse H, Vermorel C, Pinsault N. Physiotherapists as first-contact practitioners for patients with low back pain in French primary care: a pragmatic cluster randomised controlled trial. BMC Health Serv Res. 2024 Nov 18;24(1):1427. doi: 10.1186/s12913-024-11814-2. PMID 39558330